CLINICAL TRIAL: NCT00652158
Title: A Phase 1 Trial of Extended MLN8054 Dosing in Patients With Advanced Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C10002
Record Dates: First submitted 2008-03-31; First posted 2008-04-03 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-09

CONDITIONS: Advanced Malignancies
MeSH Terms: interventions — MLN8054

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: MLN8054

INTERVENTIONS:
Drug: MLN8054 — 10 mg doses of MLN8054 were given orally once daily following a schedule of "5 days on/2 days off/5 days on" repeated every 28 days

SUMMARY:
This is a phase 1 clinical trial designed to evaluate increasing durations of MLN8054 oral dosing in patients with advanced malignancies. MLN8054 will be given once daily for 4 to 7 consecutive days per week for 2 to 3 weeks. Following the 2- to 3-week treatment period there will be a 2 week recovery period.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following inclusion criteria to be enrolled in the study:

* Has a histologically or cytologically confirmed metastatic and/or advanced malignancy (including lymphomas but excluding malignancies with extensive bone marrow involvement such as leukemias and multiple myeloma) for which standard treatment does not offer curative or life-prolonging potential
* Aged 18 years or more
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Expected survival longer than 3 months from enrollment in the study
* Radiographically or clinically evaluable tumor; however, measurable disease is not required for participation in this study
* Suitable venous access for the conduct of blood sampling for determination of MLN8054 plasma concentrations
* Willingness to have serial skin punch biopsies obtained and, if feasible, to have serial biopsies of tumor tissue obtained before and following the first dose of MLN8054 Note: Once the relationship between drug exposure and inhibition of Aurora A kinase activity has been established, patients subsequently enrolled in the study will not be required to undergo either tumor or skin biopsies.

  8. Recovered from the reversible effects of prior antineoplastic therapy with at least 4 weeks elapsed since the last exposure to cytotoxic chemotherapy or radiotherapy and at least 6 weeks elapsed since exposure to nitrosoureas or mitomycin C. Patients treated with fully human monoclonal antibodies must not have received treatment with such antibodies for at least 6 weeks, and those treated with chimeric monoclonal antibodies must not have received treatment with such antibodies for at least 4 weeks. Patients treated with noncytotoxic small molecule drugs (eg, tyrosine kinase inhibitors such as Tarceva and hormonal agents such as Femara®) must not have received treatment with these drugs for at least 2 weeks before the first dose of MLN8054 is given.
* Male patients must use an appropriate method of barrier contraception (ie, condoms) and inform any sexual partner that she must also use a reliable method of contraception (eg, a hormonal contraceptive, an intrauterine device, or diaphragm with spermicide) during the study and for 3 months after the last dose of study treatment.
* Female patients must be postmenopausal, surgically sterilized, or willing to use reliable methods of birth control (eg, a hormonal contraceptive, an intrauterine device, diaphragm with spermicide, or abstinence) during the study and for 3 months after the last dose of study treatment. They should inform any male sexual partner to use an appropriate method of barrier contraception (ie, condoms) as well.
* Able to give informed consent before the conduct of any study-related procedure not part of normal medical care and able to comply with the protocol

Exclusion Criteria:

Patients meeting any of the following exclusion criteria are not to be enrolled in the study:

* Pregnant or lactating
* Major surgery within the 21 days preceding the first dose of study treatment
* Infection requiring antibiotic therapy within the 7 days preceding the first dose of study treatment
* Life-threatening illness unrelated to cancer
* Ongoing nausea or vomiting greater than Grade 1 in severity. Patients who require ongoing treatment with metoclopramide to control nausea or vomiting, to the point that it is Grade 1 or less in severity, are allowed to participate in this trial.
* Diarrhea greater than Grade 1 in severity. Patients who require ongoing therapy with an antimotility agent to control diarrhea to a Grade 1 or lower level are not allowed to participate in this trial.
* Known GI disease that could interfere with the oral absorption or tolerance of MLN8054
* Difficulty swallowing capsules
* Inability to remain nothing by mouth (NPO), except for water and prescribed medications, for 2 hours preceding and 2 hours following each dose of MLN8054
* Received more than 4 previous cytotoxic chemotherapeutic regimens including regimens used as adjuvant or neo-adjuvant therapies. There is no limit on the number of noncytotoxic therapies (eg, hormonal and immunologic) that patients may have received. Tyrosine kinase inhibitors (eg, Tarceva and Iressa®) are considered noncytotoxic compounds.
* Prior treatment with high-dose chemotherapy, defined as chemotherapy requiring the use of peripheral blood or bone marrow stem cell support for hematopoietic reconstitution
* Prior treatment with radiation therapy involving greater than or equal to 25% of the hematopoietically active bone marrow
* Clinical and/or radiographic evidence of cerebral metastases. However, patients who have a history of CNS metastasis but have no radiographic or clinical evidence of residual tumor (eg, following complete surgical resection) are not excluded from participation in this study.
* Absolute neutrophil count <1.5 x 106/ul; platelet count <100 x 106/ul.
* Serum creatinine >1.6 mg/dL or a measured or estimated (Cockcroft-Gault formula) creatinine clearance <30 mL/minute
* Bilirubin >1.25 times the upper limit of the normal range (ULN); aspartate aminotransferase (AST)/alanine aminotransferase (ALT) >2 times the ULN, and alkaline phosphatase (ALP) >2 times the ULN. Both the AST and ALP may be elevated up to 5 times the ULN if their elevation can be reasonably ascribed to the presence of metastatic disease to liver and/or to bone; however, the ALT must in all circumstances be <2 times the ULN.
* Abnormalities or arrhythmias on 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, are considered to be clinically significant
* Known or suspected human immunodeficiency virus (HIV) positive or hepatitis B surface antigen-positive status or known or suspected active hepatitis C infection
* Known or suspected disorder of bilirubin metabolism or excretion including, but not limited to, Gilbert's syndrome, Crigler-Najjar syndrome, Dubin-Johnson syndrome, and Rotor syndrome
* Inclusion in a trial of an investigational drug in the previous 4 weeks
* Admission of alcohol abuse or an inability to restrict consumption of alcohol to no more than 1 standard unit of alcohol per day during the study and for 21 days from the last dose of study treatment. A standard unit of alcohol is defined as one 12 oz beer, 1.5 oz of 80 proof alcohol, or one 6 oz glass of wine.

Note: criteria 22, 23, and 24 apply only to patients in whom biopsy of tumor tissue is planned.

* aPTT and/or PT exceeding the ULN
* Known bleeding diathesis or history of abnormal bleeding
* Ongoing therapy with an anticoagulant (eg, aspirin, plavix, coumadin, heparin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2006-04; Primary Completion 2008-03 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Toxicities of MLN8054 therapy will be identified by continuous monitoring of adverse events, by at least once weekly assessment of laboratory values (hematology and clinical chemistry),and by periodic physical examinations and vital sign measurements | 12 - 18 months

SECONDARY OUTCOMES:
Serial physical examinations, blood samples for tumor marker measurements, and radiographic evaluations will be used to assess the status of the patient's underlying disease | completion of every 2 cycles of MLN8054 treatment using theRECIST guidelines

CONTACTS AND LOCATIONS:
Locations (1):
- Ciutat Sanitaria Vall d'Hebron, Barcelona, Spain